CLINICAL TRIAL: NCT06490276
Title: Effects of Biofeedback Gait Training on Gait Quality Post-stroke
Brief Title: Biofeedback Gait Training on Gait Quality in Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yea-Ru Yang, Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NYCU112205AF2
Record Dates: First submitted 2024-06-30; First posted 2024-07-08 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Stroke
Keywords: Biofeedback; Gait symmetry; Gait variability; Gait training
MeSH Terms: conditions — Stroke | interventions — Biofeedback, Psychology

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gait training with biofeedback group (Experimental): The intervention is a 60-minute session and 3 sessions/week, totaling 4 weeks.
  Interventions: Other: Gait training with biofeedback
- Gait training without biofeedback group (Active Comparator): The intervention is a 60-minute session and 3 sessions/week, totaling 4 weeks.
  Interventions: Other: Gait training without biofeedback

INTERVENTIONS:
Other: Gait training with biofeedback — Gait training include treadmill and overground walking. The biofeedback device system will provide real-time feedback on hip extension angles.
  Arms: Gait training with biofeedback group
Other: Gait training without biofeedback — Gait training include treadmill and overground walking.
  Arms: Gait training without biofeedback group

SUMMARY:
Post-stroke gait dysfunction is characterized by reduced gait velocity and stride length, along with gait asymmetry and instability. Gait asymmetry and instability are considered as indicators for gait quality, which affect independence and quality of life in individual with stroke. Previous studies have suggested that gait biofeedback is a promising strategy for enhancing the efficacy of post-stroke gait training. However, there is insufficient evidence on the effects of kinematic biofeedback gait training on gait asymmetry and instability in individuals with stroke. Therefore, the purpose of this study is to investigate the effects of real-time kinematic gait biofeedback training on gait quality in individuals with stroke.

ELIGIBILITY:
Inclusion Criteria:

* First stroke
* Stroke onset time ≥ 6 months
* Functional Ambulation Category ≥3
* Passive range of motion of affected hip extension is at least 10 degrees
* Mini-Mental State Measurement score ≥ 24 points

Exclusion Criteria:

* Modified Ashworth Scale of affected ankle plantar flexors ≥ 2
* Muscle strength of affected ankle plantar flexors via Manual Muscle Testing ≤ 1
* Uncorrected auditory impairment
* Severe cardiovascular disease or uncontrolled hypertension
* Other orthopedic diseases that may affect walking ability
* Other neurological disease except stroke

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Gait symmetry | Change from baseline at 4 weeks after training and 4 weeks follow-up
  Using GAITRite system to measure the symmetry of saptiotemporal parameters
Gait variability | Change from baseline at 4 weeks after training and 4 weeks follow-up
  Using GAITRite system to measure the coefficient of variation of saptiotemporal parameters

SECONDARY OUTCOMES:
Propulsive force | Change from baseline at 4 weeks after training and 4 weeks follow-up
  Using Force plate to measure the ground reaction force
Gait performance | Change from baseline at 4 weeks after training and 4 weeks follow-up
  Using the GAITRite system to evaluate saptiotemporal parameters
Berg Balance Scale | Change from baseline at 4 weeks after training and 4 weeks follow-up
  Using Berg Balance Scale to evaluate balance ability
Activities-specific Balance Confidence Scale | Change from baseline at 4 weeks after training and 4 weeks follow-up
  Using Activities-specific Balance Confidence Scale to evaluate individual's balance confidence in performing daily activities
Taiwan Chinese version Falls Efficacy Scale | Change from baseline at 4 weeks after training and 4 weeks follow-up
  Using Taiwan Chinese version Falls Efficacy Scale to evaluate concerns about falling
Frenchay Activities Index | Change from baseline at 4 weeks after training and 4 weeks follow-up
  Using Frenchay Activities Index to measure individual's capacity to perform instrumental activities of daily living
Stroke Impact Scale | Change from baseline at 4 weeks after training and 4 weeks follow-up
  Using Stroke Impact Scale to evaluate disability and quality of life after stroke

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Therapy and Assistive Technology, National Yang Ming Chiao Tung University, Taipei, Taiwan